CLINICAL TRIAL: NCT04216810
Title: The Effectiveness of Adding Cupping Therapy in Patients With Nonspecific Chronic Lumbar Pain: a Randomized Controlled Study.
Brief Title: The Effectiveness of Adding Cupping Therapy in Patients With Nonspecific Chronic Lumbar Pain
Acronym: lowbackpain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sidnei Correia
Record Dates: First submitted 2019-12-26; First posted 2020-01-03 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Low Back Pain, Mechanical; Low Back Pain, Postural; Lower Back Pain Chronic; Low Back Pain, Posterior Compartment
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Active Comparator): Exercise group
  Interventions: Other: muscle strengthening exercises
- Exercise group and dry cupping (Experimental): Exercise and dry cupping
  Interventions: Other: muscle strengthening exercises and dry cupping

INTERVENTIONS:
Other: muscle strengthening exercises — segmental stabilization exercises
  Arms: Exercise group
Other: muscle strengthening exercises and dry cupping — segmental stabilization exercises and dry cupping
  Arms: Exercise group and dry cupping

SUMMARY:
Low back pain is a major public health problem and is associated with a high rate of absenteeism at work, functional disability and frequent use of health services. Suction cup therapy is a common technique of traditional Chinese medicine (TCM), which has been around for about 3,300 years in Asia and the Middle East and has as its main feature the decrease in signs and symptoms of chronic pain. The technique was widely used in the 19th century throughout Asia and Europe, and in recent years demand has been increasing, possibly due to the inefficiency of conventional therapies and medicines. Objective: To verify the effectiveness of the suction cup therapy technique associated with conventional physiotherapy in patients with chronic low back pain. Method: We will include individuals between 18 and 60 years old, both genders, with low back pain for more than 3 months, without having received physical therapy treatment for a period of 6 months. Individuals with severe spinal diseases, root conditions of the spine, carriers of vascular diseases and pregnant women will be excluded. They will be randomly divided into two groups, Conventional Physiotherapy (group 1) and Conventional Physiotherapy associated with suction cup therapy (group 2).

ELIGIBILITY:
Inclusion Criteria:

* nonspecific chronic low back pain without lower limb irradiation
* Aged between 18 and 60 years,
* Both genders
* Low back pain for more than 3 months
* Without having received physiotherapy treatment for a period of 6 months

Exclusion Criteria:

* individuals with severe spinal diseases (fractures, tumors and inflammatory conditions such as ankylosing spondylitis)
* root conditions of the spine (disc herniation and spondylolisthesis with neurological impairment and narrowing of the spinal canal)
* root conditions of the spine
* carriers of vascular diseases
* pregnant women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
pain intensity after and before six weeks | immediately after the intervention
  Numerical Visual Scale (0-100)

CONTACTS AND LOCATIONS:
Locations (1):
- Claudio Cazarini Júnior, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Walker BF. The prevalence of low back pain: a systematic review of the literature from 1966 to 1998. J Spinal Disord. 2000 Jun;13(3):205-17. doi: 10.1097/00002517-200006000-00003. PMID 10872758
- [Result] Dagenais S, Caro J, Haldeman S. A systematic review of low back pain cost of illness studies in the United States and internationally. Spine J. 2008 Jan-Feb;8(1):8-20. doi: 10.1016/j.spinee.2007.10.005. PMID 18164449
- [Result] Dagenais S, Roffey DM, Wai EK, Haldeman S, Caro J. Can cost utility evaluations inform decision making about interventions for low back pain? Spine J. 2009 Nov;9(11):944-57. doi: 10.1016/j.spinee.2009.07.007. Epub 2009 Sep 12. PMID 19748833
- [Result] Areeudomwong P, Buttagat V. Proprioceptive neuromuscular facilitation training improves pain-related and balance outcomes in working-age patients with chronic low back pain: a randomized controlled trial. Braz J Phys Ther. 2019 Sep-Oct;23(5):428-436. doi: 10.1016/j.bjpt.2018.10.005. Epub 2018 Oct 17. PMID 30361077